CLINICAL TRIAL: NCT07399249
Title: Usability and Clinical Validation of the NowFuture Digital Flu / COVID Test in Anterior Nasal Samples for Over-The-Counter (OTC) Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocrucible Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLN-0019; 75A50125C00003 (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority (BARDA))
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: SARS CoV 2 Infection; Influenza A Virus Infection; Influenza B Virus Infection
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): Participants self-collecting and testing the device themselves or collecting a sample and performing the testing on another participant
  Interventions: Diagnostic Test: Diagnostic test for SARS-CoV-2, influenza A and influenza B

INTERVENTIONS:
Diagnostic Test: Diagnostic test for SARS-CoV-2, influenza A and influenza B — Participants will test themselves or another participant for SARS-CoV-2, influenza A and influenza B. Participants will observe the test result displayed on the device. Participants will be advised to not use investigational test result for diagnostics purposes.

SUMMARY:
Prospective clinical study conducted at three or more geographically diverse sites (with a simulated home environment) in the United States for the clinical validation of the NowFuture Digital Flu / COVID Test. Results from the investigational test will be compared to results from a 510(k) cleared highly sensitive reverse transcriptase polymerase chain reaction (RT-PCR) test for SARS-CoV-2, Influenza A and Influenza B. The primary objective of this study is to evaluate the clinical performance (positive percent agreement, negative percent agreement and 95% confidence intervals for upper and lower bounds) of the NowFuture Digital Flu / COVID Test for the qualitative detection and differentiation of SARS-CoV-2 nucleocapsid antigen, Influenza A and Influenza B nucleoproteins antigens using AN swab samples collected and processed in the test by lay users. The secondary objective is to evaluate the usability of the investigational test and the user comprehension of the investigational test lay user instructions when performed by the lay users.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to study enrollment.
* Male or female aged 2 years of age and older.
* Participant is currently exhibiting at least one symptom (i.e. symptomatic) associated with COVID-19 or influenza (such as, but not limited to, fever, headache, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea) and must present within 6 days of symptom onset (equates to 5 DPSO). Subject must still be exhibiting symptom(s) on the day of sample collection.

Exclusion Criteria:

* Participant or participant's legally acceptable representative (for minors) who is 18 years of age (or the state's legal age of majority) or older and does not understand or is not able and willing to sign the study informed consent.
* Participant who has had a positive SARS-CoV-2, Influenza A and/or Influenza B result within the past 30 days.
* Participant has had seasonal influenza vaccine such as the FluMist/FluMist Quadrivalent live intranasal influenza vaccine and/or the SARS-CoV-2 vaccine within the past 5 days.
* Participant is not able to tolerate sample collection or is not willing to contribute the required swab samples for testing or complete the study procedures.
* Participant is currently undergoing antiviral treatment such as baloxavir marboxil (Xofluza), oseltamivir (Tamiflu®), zanamivir (Relenza®), and peramivir (Rapivab®).
* Participant currently undergoing treatment and/or has undergone treatment within the past thirty (30) days with prescription medication to treat Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury), Paxlovid, molnupiravir or receiving convalescent plasma therapy for SARS-CoV-2.
* Participant who has had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to the study sample collection.
* Participant who has had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | The duration from enrollment to ending participation is one day. Each test session is estimated to last 60 minutes and conclude following test and comparator sample collection and completion of participant questionnaire.
  Clinical performance (positive percent agreement, negative percent agreement and 95% confidence intervals for upper and lower bounds) of the NowFuture Digital Flu / COVID Test for the qualitative detection and differentiation of SARS-CoV-2 nucleocapsid antigen, Influenza A and Influenza B nucleoproteins antigens using AN swab samples collected and processed in the test by lay users and compared to results from a 510(k) cleared highly sensitive reverse transcriptase polymerase chain reaction (RT-PCR) test for SARS-CoV-2, influenza A and influenza B. The primary outcome of the study requires a minimum of; 50 SARS-CoV-2 positive samples, 50 Influenza A positive samples, 30 Influenza B positive samples and 500 negative samples by comparator. Study must be performed within a US Flu season, i.e. October to April of any given year.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2026-01-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT07399249/ICF_000.pdf